CLINICAL TRIAL: NCT04225065
Title: Does Chlorhexidine and/or Betadine Prep Thoroughly Clean the Surgical Sites and Fingernails in Pediatric Arm Surgery Following Trauma?
Brief Title: Chlorhexidine and/or Betadine Prep in Pediatric Arm Surgery Following Trauma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI does not wish to proceed with study.
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-0106
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Arm Fracture; Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Chlorhexidine; Povidone-Iodine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Chlorhexidine prep (Active Comparator): Chlorhexidine prep prior to their operation
  Interventions: Other: Chlorhexidine
- Betadine prep (Active Comparator): Betadine prep prior to their operation
  Interventions: Other: Betadine

INTERVENTIONS:
Other: Chlorhexidine — Chlorhexidine prep prior to surgery
  Arms: Chlorhexidine prep
Other: Betadine — Betadine prep prior to surgery
  Arms: Betadine prep

SUMMARY:
There have been numerous studies demonstrating surgical site infections that arise from contamination at time of surgery or by seeding from other sites in the body which arise from organisms normally found on the skin. This has been known to cause complications in spine surgery, shoulder, hip, and knee arthroplasty. While studies have shown that organisms like Cutibacterium persists on the skin despite standard surgical preparation, there have not been studies that examine the organisms found in the fingernail region pre- and post- standard surgical preparations. This study investigates how thorough fingernails are prepped prior to the operation. The results of this study would determine whether providers are adequately cleaning the patient's entire arm, including under the fingernail, prior to surgery. The results may support continuation of the current practice or adding to the standard surgical preparation to ensure adequately sterilization of surgical sites and all exposed areas, which include the fingernails.

DETAILED DESCRIPTION:
It is well known that even with surgical skin preparation, there are some microorganisms that remain on the patient's skin. There have been numerous studies demonstrating surgical site infections that arise from contamination at time of surgery or by seeding from other sites in the body which arise from organisms normally found on the skin. This has been known to cause complications in spine surgery, shoulder, hip, and knee arthroplasty. While studies have shown that organisms like Cutibacterium persist on the skin despite standard surgical preparation, there have not been studies that examine the organisms found in the fingernail region pre- and post- standard surgical preparations. It is common practice to not cover the fingernails when patients are undergoing distal upper extremity surgery. Providers tend to consider them prepped when they have the chlorhexidine or betadine preparations applied; however, there is uncertainty regarding how much attention is given to the fingernails. This study investigates how thorough fingernails are prepped prior to the operation. The results of this study would determine whether providers are adequately cleaning the patient's entire arm, including under the fingernail, prior to surgery. The results may support continuation of the current practice or adding to the standard surgical preparation to ensure adequate sterilization of surgical sites and all exposed areas, which include the fingernails.

This is a prospective study design of 20 pediatric patients who are undergoing distal upper extremity surgery. Ten patients will receive a chlorhexidine prep prior to their operation, and the other 10 will receive a betadine prep. Patients will be considered for the study if they are 10 years old or younger and are having either wrist, forearm, or elbow internal fixation surgeries. Three culture specimens will be sent to microbiology: 1) before the surgical skin preparation; 2) after the skin preparation but before the operation; and 3) after the operation. Culture results will be compared pre- and post- surgical prep and between chlorhexidine and betadine preps.

ELIGIBILITY:
Inclusion Criteria:

* Patient less than or equal to 10 years of age
* Undergoing wrist, forearm, or elbow internal fixation surgery

Exclusion Criteria:

* Patient with known immunodeficiency disorder

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Type and number of organisms found in culture | 1 day
  Type and number of organisms found in fingernail culture

CONTACTS AND LOCATIONS:
Overall Officials: Mark Seeley, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Woodbine, Danville, Pennsylvania, United States